CLINICAL TRIAL: NCT01845324
Title: Relation Between Fetal Heart Interventricular Septum Size and Gestational Diabetes Mellitus Control. a Prospective Trial
Brief Title: Fetal Heart Interventricular Septum in Fetuses of Diabetic Mothers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0011-13
Record Dates: First submitted 2013-04-09; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Pregnancy; Diabetes Mellitus
Keywords: Pregnancy; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes Mellitus in pregnancy: Our cohort will include all consequtive women with Diabetes Mellitus atending our clinic

SUMMARY:
The investigators asume that the measurement of the fetal heart interventricular septum can serve as a good tool to predict glucose control in pregnant patients with diabetes mellitus. The investigators will measure the septum width in patients with Diabetes and will correlate to standard measurements of the glucuse levels.

DETAILED DESCRIPTION:
In this study the investigators will follow patients with Diabetes Mellitus - mainly gestational. the investigators will measure the width of the interventricular septum and correlate with conventional measures of blood glucose measurements in this population.

The investigators will try to assess whether measurement of the septum can be an earlier and better predictor of glucose control in this population.

ELIGIBILITY:
Inclusion Criteria:

* All consequtive pregnant women
* with Diabetes Mellitus - Gestational and non Gestational

Exclusion Criteria:

.No willing to participate.

* Suspected Heart anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All consequtive pregnant women with Diabetes Mellitus - Gestational and non Gestational
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
width of fetal interventricula heart septum | 2 years
  The investigator will assess the width of the fetal interventricular septum in patients with diabetes.

SECONDARY OUTCOMES:
glucose control in patients with normal and abnormal interventricular septal width | 2 years
  The investigators will try to show that small interventricular septal width glucose correlates with good glucose control

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel